CLINICAL TRIAL: NCT07393776
Title: Effects of a Semantically Irrelevant Virtual Reality Experience on Memory and Emotion After Watching a Traumatic Event: Randomized Controlled Experimental Study
Brief Title: Effects of Semantically Irrelevant Virtual Reality Experience on Memory and Emotion
Acronym: FIRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-966
Record Dates: First submitted 2026-01-09; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Intervention Group; Comparison Group; Control Group
Keywords: virtual reality; mental health; memory suppression; emotion
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: In stage 1, participants in all groups watched a short video of an actual severe house fire to create a traumatic event memory. In stage 2, the control group stayed seated without doing anything, the comparison group read a paragraph about the Egyptian Ocean as semantically irrelevant follow-up information, and the intervention group watched a 360° VR video of the Egyptian Ocean that features opposite attributes to the fire (eg, blue water vs red fire, cool water vs hot fire).
Who Masked: Participant
Masking Description: Participants were masked about the group they were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group (Active Comparator): Intervention Group participants watched semantically irrelevant VR video of the Red Sea underwater diving 5 minutes after participants watched the fire video.
  Interventions: Other: Watching VR video
- Control (No Intervention): Control group participants did not receive any intervention.
- Comparison Group (Placebo Comparator): Comparison Group participants read text description of the Red Sea underwater diving 5 minutes after participants watched the fire video.
  Interventions: Other: Reading text

INTERVENTIONS:
Other: Watching VR video — Participants watch 360-degree VR video of underwater diving 5 minutes after they watched the fire video.
  Arms: Intervention Group
Other: Reading text — Participants read text paragraphs regarding underwater diving 5 minutes after they watched the fire video.
  Arms: Comparison Group

SUMMARY:
First responders at the Federal, State and local level are those on the front lines of providing support to their communities during an emergency or a disaster. Their work domains are emergency public security, firefighting, law enforcement, emergency response, and emergency medical care. Due to the inherent characteristics of the jobs they perform, they are constantly exposed to very stressful, demanding and dangerous work environments. Such an exposure often leads to mental health issues such as anxiety, depression, and post-traumatic stress disorder (PTSD). More than 80 percent of first responders experience traumatic events on their job duty. Various efforts to treat about trauma have been made to address the first responders' mental health. However, existing interventions are not directly targeted at the causes of mental health problems, which is the memory of the adverse events. The objective the proposed research is to investigate the effect of immersive virtual reality (VR) experience on the memory of an adverse event (e.g., fire).

DETAILED DESCRIPTION:
Background: First responders, such as firefighters, experience significant mental health issues due to the high-stress nature of their work. Existing mental health interventions, such as meditation and debriefing, despite their benefits, do not target cognitive processing of traumatic events such as memory and emotion.

Objective: This work aims to examine effects of semantically irrelevant virtual reality (VR) content to intervene in the retrieval of an adverse event memory and its associated emotions. Cognitive models of posttraumatic stress disorder posit that exposure to stimuli that are similar to a previous trauma acts as a trigger for retrieval of the associated memory and bodily reaction (eg, elevated heart rate). This work uses semantically irrelevant VR as an intervention to interrupt the retrieval of the traumatic memory by placing a participant in a VR environment that has a distant semantic connection to the trauma.

Methods: A total of 107 participants recruited from a large public university in Texas was randomly assigned to 1 of 3 groups: control (n=33), comparison (n=37), and intervention (n=37). In stage 1, participants in all groups watched a short video of an actual severe house fire to create a traumatic event memory. In stage 2, the control group stayed seated without doing anything, the comparison group read a paragraph about the Egyptian Ocean as semantically irrelevant follow-up information, and the intervention group watched a 360° VR video of the Egyptian Ocean that features opposite attributes to the fire (eg, blue water vs red fire, cool water vs hot fire). The Positive and Negative Affect Schedule, which has 10 items for positive emotions (eg, attentive and excited) and 10 items for negative emotions (eg, scared and distressed), was administered after each of the two stages. In stage 3, the memory accuracy of the house fire video was assessed using a forced recognition test of 15 pairs of a true image and a fake image generated by artificial intelligence software.

ELIGIBILITY:
Inclusion Criteria:

* aged at least 18 years
* currently enrolled at the university

Exclusion Criteria:

* under 18 years
* not currently enrolled at the university

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Memory accuracy | Immediately after participants received the intervention.
  The ratio of correct images participants chose from two images of the fire video they watched.

SECONDARY OUTCOMES:
Positive And Negative Affect Schedule (PANAS) | Immediately after participants watched the fire video and immediately after they watched the VR video (intervention) or read the text (comparison).
  PANAS consists of 10 positive affects and 10 negative affects each with a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Changwon Son, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Industrial, Manufacturing, & Systems Engineering Department, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Son, C., Parker, K., & Jamshidzadeh, M. (2026). Effects of a Semantically Irrelevant Virtual Reality Experience on Memory and Emotion After Watching a Traumatic Event: Randomized Controlled Experimental Study. JMIR Formative Research